CLINICAL TRIAL: NCT02739009
Title: First in Human of Single and Multiple Doses of MOR106
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Collaborators: MorphoSys AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MOR106-CL-101
Record Dates: First submitted 2016-04-01; First posted 2016-04-14 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Healthy; Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- MOR106 (Experimental): Single intravenous administration of MOR106
  Interventions: Drug: MOR106 single ascending doses, intravenous
- Placebo (Placebo Comparator): Single intravenous administration of Placebo
  Interventions: Drug: Placebo single ascending doses, intravenous
- MOR106 MAD (Experimental): Multiple intravenous administration of MOR106
  Interventions: Drug: MOR106 multiple ascending doses, intravenous
- Placebo MAD (Placebo Comparator): Multiple intravenous adminstration of Placebo
  Interventions: Drug: Placebo multiple intravenous administrations

INTERVENTIONS:
Drug: MOR106 single ascending doses, intravenous
  Arms: MOR106
Drug: Placebo single ascending doses, intravenous
  Arms: Placebo
Drug: MOR106 multiple ascending doses, intravenous
  Arms: MOR106 MAD
Drug: Placebo multiple intravenous administrations
  Arms: Placebo MAD

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose-escalation, phase I study for the assessment of safety, tolerability and pharmacokinetics of single ascending doses of MOR106 in healthy male subjects and multiple ascending doses in subjects with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

- Able and willing to give voluntary written informed consent

Single ascending dose (SAD)

* Negative urine drug screen
* Male between 18-50 years of age
* A body mass index (BMI) between 18-30 kg/m², inclusive.
* Judged to be in good health

Multiple ascending dose (MAD)

* Male or female between 18-65 years of age
* A BMI between 18-30 kg/m²
* Diagnosis of Atopic Dermatitis (AD) for at least 6 months as per the Hanifin and Rajka Criteria
* EASI ≥ 16 at the screening and baseline visits
* IGA score ≥3 (on the 0 to 4 IGA scale, in which 3 is moderate and 4 is severe) at the screening and baseline visits
* Greater than or equal to 10% body surface area (BSA) of AD involvement at screening
* Willingness to continue stable use of an additive free, basic, bland emollient twice daily for at least 7 days before the baseline visit
* Subject is a candidate for systemic therapy and is not responding adequately or has a contraindication to topical corticosteroids and/or topical calcineurin inhibitors (per Investigator's judgement)
* Absence of current active, latent or history of tuberculosis (TB) infection based on medical history and as determined by a negative QuantiFERON TB Gold test at screening
* Female subjects must have a negative serum pregnancy test at screening and a negative urine pregnancy test at baseline
* Female subjects of childbearing potential must use a highly effective method contraception from 28 days prior to the first dose of study drug, during the study and for at least 24 weeks after the last dose

Exclusion Criteria:

* Known hypersensitivity to study drug ingredients.
* History of or a current immunosuppressive condition
* Symptoms of clinically significant illness in the 3 months before the initial study drug administration.
* Any concurrent illness, condition, disability, or clinically significant abnormality
* Treatment with any drug known to have a well-defined potential for toxicity to a major organ in the last 3 months preceding the initial study drug administration.
* A history of significant psychological, neurologic, hepatic, renal, endocrine, cardiovascular, gastrointestinal (GI), pulmonary, or metabolic disease.

MAD only

* Active (skin) infection requiring systemic antibiotics
* immunosuppressive/immunomodulating drugs or phototherapy 4 weeks prior to baseline
* Treatment with topical corticosteroids (TCS) or topical calcineurin inhibitors (TCI) within 2 weeks before the baseline
* Treatment with biologics within 5 half-lives (if known) or 12 weeks prior to baseline visit
* history of immunosuppression
* Regular use (more than 2 visits per week) of a tanning booth/ parlor within 4 weeks of the screening visit
* Regular daily use of oral nonsteroidal anti-inflammatory drugs (NSAIDs), except low-dose aspirin (≤200 mg/day) for cardioprotection, within 7 days prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-04; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Difference as compared to placebo in the number of subjects with treatment-emergent adverse events | Up to 99 days after dosing
  To evaluate the safety and tolerability of single ascending doses of MOR106 intravenously given to healthy male subjects and of multiple ascending doses of MOR106 given intravenously to subjects with atopic dermatitis, compared to placebo
Difference as compared to placebo in the number of subjects with deviating physical examination results | Up to 99 days after dosing
  To evaluate the safety and tolerability of single ascending doses of MOR106 intravenously given to healthy male subjects and of multiple ascending doses of MOR106 given intravenously to subjects with atopic dermatitis, compared to placebo
Difference as compared to placebo in the number of subjects with abnormal vital signs | Up to 99 days after dosing
  To evaluate the safety and tolerability of single ascending doses of MOR106 intravenously given to healthy male subjects and of multiple ascending doses of MOR106 given intravenously to subjects with atopic dermatitis, compared to placebo
Difference as compared to placebo in the number of subjects with abnormal 12-lead ECG results | Up to 99 days after dosing
  To evaluate the safety and tolerability of single ascending doses of MOR106 intravenously given to healthy male subjects and of multiple ascending doses of MOR106 given intravenously to subjects with atopic dermatitis, compared to placebo
Difference as compared to placebo in the number of subjects with abnormal laboratory findings | Up to 99 days after dosing
  To evaluate the safety and tolerability of single ascending doses of MOR106 intravenously given to healthy male subjects and of multiple ascending doses of MOR106 given intravenously to subjects with atopic dermatitis, compared to placebo
Difference as compared to placebo in the occurrence of infusion related reactions | Up to 99 days after dosing
  To evaluate the safety and tolerability of single ascending doses of MOR106 intravenously given to healthy male subjects and of multiple ascending doses of MOR106 given intravenously to subjects with atopic dermatitis, compared to placebo

SECONDARY OUTCOMES:
Serum concentration (Cinf) of MOR106 | up to 99 days after dosing
  To characterize the PK of MOR106 after single intravenous administration in healthy male volunteers and after multiple ascending dose intravenous administration in subjects with severe atopic dermatitis
Area under the curve (AUC) of MOR106 | up to 99 days after dosing
  To characterize the PK of MOR106 after single intravenous administration in healthy male volunteers and after multiple ascending dose intravenous administration in subjects with severe atopic dermatitis
terminal elimination half-life (t1/2) of MOR106 | up to 99 days after dosing
  To characterize the PK of MOR106 after single intravenous administration in healthy male volunteers and after multiple ascending dose intravenous administration in subjects with severe atopic dermatitis
total serum clearance (CL) of MOR106 | up to 99 days after dosing
  To characterize the PK of MOR106 after single intravenous administration in healthy male volunteers and after multiple ascending dose intravenous administration in subjects with severe atopic dermatitis
volume of distribution at steady state (Vss) of MOR106 | up to 99 days after dosing
  To characterize the PK of MOR106 after single intravenous administration in healthy male volunteers and after multiple ascending dose intravenous administration in subjects with severe atopic dermatitis
The presence of anti-drug antibodies in serum over time after single intravenous dose | up to 9 days after dosing
  To assess the presence of anti-drug antibodies as a measure of immunogenicity after single administration of MOR106 and after multiple ascending dose intravenous administration in subjects with severe atopic dermatitis

CONTACTS AND LOCATIONS:
Overall Officials: Helen Timmis, MBChB, Study Director — Galapagos NV
Locations (4):
- SGS LSS Clinical Pharmacology Unit, Antwerp, Belgium
- St Johns Hospital, Budapest, Hungary
- • Arensia Phase I unit, Chisinau, Moldova
- Arensia Phase I unit, Bucharest, Romania